CLINICAL TRIAL: NCT04305691
Title: A Phase 2 Trial of Ixazomib for Kaposi Sarcoma
Brief Title: Trial of Ixazomib for Kaposi Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-107; NCI-2020-01138 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-107 (Other: AIDS Malignancy Consortium); AMC-107 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Kaposi Sarcoma; Skin
Keywords: Kaposi Sarcoma; HIV; Skin; ixazomib
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (ixazomib) (Experimental): Patients receive ixazomib PO on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response may continue treatment for an additional 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib Citrate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ixazomib works in treating patients with Kaposi sarcoma. Ixazomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the overall response rate of ixazomib in participants with Kaposi sarcoma.

SECONDARY OBJECTIVES:

I. Determine safety and tolerability of ixazomib. II. Assess changes in Kaposi-sarcoma associated herpesvirus (KSHV) viral load (VL) by ixazomib.

III. Correlate changes in KSHV VL with tumor response. IV. For human immunodeficiency virus (HIV)-positive participants, assess changes in CD4 counts and HIV viral load.

EXPLORATORY OBJECTIVE:

I. Assess changes in quality of life during ixazomib therapy.

OUTLINE:

Patients receive ixazomib orally (PO) on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response may continue treatment for an additional 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks, then periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participants must have histologically or cytologically confirmed cutaneous Kaposi sarcoma. Participants must have measurable disease with a minimum of five bi-dimensionally measurable KS cutaneous marker lesions. If fewer than five bi-dimensionally measurable marker lesions are available, the total surface area of the marker lesion(s) must be >= 700 mm^2
* Participants must have documentation of HIV status. If HIV negative, documentation of a negative HIV rapid test within 21 days before enrollment. If HIV positive, documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care provider
  * Documentation of receipt of antiretroviral therapy (ART) (at least two different medications that do not constitute a prescription for pre exposure prophylaxis [PrEP]) by a licensed health care provider. Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating > 1000 RNA copies/mL
  * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or Multispot HIV-1/HIV-2 Rapid Test or HIV Antibody HIV-1/HIV-2 Differentiation Assay

    * Note: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally (e.g., United States [U.S.] Food and Drug Administration [FDA]). WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an extracellular interactome assay (E/CIA )that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count: >= 1,000/mm^3 (within 21 days before enrollment)
* Hemoglobin: > 8 g/dL (within 21 days before enrollment)
* Platelets: >= 75,000/mm^3 (within 21 days before enrollment). Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN) (within 21 days before enrollment)

  * If the elevated bilirubin is felt to be secondary to indinavir or atazanavir therapy, then subjects will be allowed on protocol without any limit on the total bilirubin if the direct bilirubin is normal
* Creatinine:

  * Serum creatinine levels within normal institutional limits; or, creatinine clearance >= 30 mL/min (as calculated per the Cockcroft-Gault Equation (within 21 days before enrollment)
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification within 6 months before study enrollment. To be eligible for this trial, participants must be class 2B or better within 6 months before enrollment
* Ixazomib can cause fetal harm. For this reason and because proteasome inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control and another method such as hormone contraception simultaneously; abstinence) before study entry, the duration of study participation, and 90 days after completion of ixazomib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception or abstain from heterosexual contact before the study, for the duration of study participation, and for 90 days after completion of ixazomib administration
* If HIV positive, participants must have been on antiretroviral therapy (ART) with optimum anti-viral response for at least 12 weeks. Three-drug ART regimens which include a protease inhibitor or a nucleoside reverse transcriptase inhibitor are acceptable, as is the recently FDA-approved injectable ART regimen, cabotegravir with rilpivirine. Additional appropriate regimens in management of HIV as specified in https://clinicalinfo.hiv.gov/ are acceptable as long as they do not include moderate or strong CYP3A4 inducers. Changes of antiretroviral therapy within the prior 12 weeks for toxicity/convenience reasons are allowed (as long as participants are on a stable regimen for 4 weeks per Section 3.1.11). However, if changes in anti-HIV therapy are due to inadequate HIV control and occurred within the 3 months prior to protocol consent, the patient is not eligible until 12 weeks after optimal control is reached.
* If HIV positive, must have been on a STABLE anti-retroviral therapy for at least 4 weeks. The non-nucleoside reverse transcriptase inhibitors (NNRTIs) efavirenz and etravirine are moderate CYP3A4 inducers which will reduce ixazomib exposure and are therefore prohibited. Potential participants requiring change of antiretroviral therapy to avoid moderate to strong CYP3A4 inducers or to pursue better HIV management with an alternate antiretroviral regimen should defer enrollment until completing 4 weeks of the new ART regimen. There should be no intention to change the regimen for the duration of the study.
* HIV positive participants must not show recent improvement in KS on ART alone that may confound response evaluation, within the following parameters:

  * If on ART 12 to 24 weeks, participants must show a burden of disease requiring further systemic KS-directed treatment (i.e. advanced cutaneous disease, presence of lymphedema or asymptomatic visceral disease, painful lesions) or evidence of KS progression:
  * i.e. any new lesion(s);
  * spreading of lesions by any measurable degree;
  * development of ulceration;
  * worsening edema documented by circumferential measure of limb or body;
  * increase in symptoms such as pain, including negative psychological impact;
  * any degree of disease worsening by imaging that would prompt expert assessment to recommend further systemic treatment with delay
  * If on ART for >24 weeks, must show no evidence of regression in last 8 weeks
* Patients who have residual active KS lesions (not merely tattoo effect) after receipt of recent KS-directed therapy are eligible to participate even if there was no interval progression since completion of therapy as long as: (1) the degree of residual disease merits systemic therapy (i.e. advanced cutaneous disease, presence of lymphedema or asymptomatic visceral disease, painful lesions)); and (2) at least 4 weeks have passed since receipt of the most recent KS-directed therapy.

Exclusion Criteria:

* Participants who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ixazomib or other agents used in study
* Chronic systemic treatment using strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort is not allowed. Patients who are on chronic use of strong CYP3A inducers must come off 14 days before receiving ixazomib treatment. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months; or psychiatric illness/social situations that would limit compliance with study requirements. This includes infections requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment but excludes ongoing antibiotic therapy for opportunistic infection (OI) prophylaxis
* Participants with a second prior or concurrent malignancy that has a natural history or treatment regimen that has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Pregnant women are excluded from this study because ixazomib is expected to cause fetal harm if used during pregnancy. It is not known if ixazomib is excreted into breast milk, but due to the potential for serious adverse events in a nursing infant, breastfeeding must be discontinued during therapy and for 90 days after the last ixazomib dose
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) before entering the study
* Participants who have not recovered from other adverse events due to prior anti-cancer therapy (i.e., have residual toxicity > grade 1), excluding alopecia
* Participants who are seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). All participants will be required to be screened for hepatitis B. Participants with resolved infection (i.e. participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc) and/or antibodies to hepatitis B surface antigen (anti-HBs) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV deoxyribonucleic acid (DNA) levels. Participants who are PCR positive will be excluded. EXCEPTION: Participants with serologic findings suggestive of hepatitis B virus (HBV) vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Participants diagnosed with hepatitis C who are hepatitis C antibody positive, whether hepatitis C RNA level is measurable or not, must have no evidence of cirrhosis and have liver function tests that conform to the protocol inclusion criteria
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Participants with grade 2 or higher peripheral neuropathy (i.e., painful neuropathy) on clinical examination during the screening period
* Major surgery within 14 days before enrollment
* Participants with symptomatic visceral Kaposi sarcoma
* Participants who have had prior treatment of Kaposi sarcoma with a proteasome inhibitor within the last 2 years or with ixazomib at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 4 weeks post treatment
  The binomial proportion and its 90% one-sided confidence interval will be used to estimate the overall response rate. Response and progression will be evaluated in this study using the acquired Immunodeficiency syndrome (AIDS) Clinical Trials Groups (ACTG) response criteria for Kaposi sarcoma, as outlined in the AIDS Malignancy Consortium (AMC) Kaposi sarcoma Response Evaluation Manual of Procedures (MOP).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 weeks post treatment
  Frequencies of toxicities will be presented by severity at the event and person level; 95% confidence intervals will be computed for the proportion of participants experiencing grade 3 and higher toxicities. The incidence of toxicity-related dose reductions and treatment discontinuations will be summarized.
Change in Kaposi-sarcoma associated herpes virus (KSHV) viral load (VL) | Baseline up to 4 weeks post treatment
  KSHV lytic gene expression over time will be summarized; changes will be graphed and explored using paired t-tests or Wilcoxon signed rank tests. KSHV levels will be correlated with tumor response by computing descriptive statistics and making exploratory comparisons according to response, as well as examining Spearman's rank correlations between tumor size KSHV levels.
Change in CD4 counts | Baseline up to 4 weeks post treatment
  Immune status over time will be summarized; changes in immune status will be graphed and explored using paired t-tests or Wilcoxon signed rank tests.
Change in human immunodeficiency virus (HIV) VL | Baseline up to 4 weeks post treatment
  HIV viral load over time will be summarized; changes in HIV VL will be graphed and explored using paired t-tests or Wilcoxon signed rank tests. HIV levels will be correlated with tumor response by computing descriptive statistics and making exploratory comparisons according to response, as well as examining Spearman's rank correlations between tumor size and HIV levels.
Complete response rate | Up to 4 weeks post treatment
  Complete response will be defined as the absence of any detectable residual disease, including tumor-associated edema, persisting for at least 4 weeks.

OTHER OUTCOMES:
Change in quality of life | Baseline up to 4 weeks post treatment
  General estimating equations will be used to evaluate changes in the functional assessment of HIV Infection (FAHI) + Kaposi sarcoma (KS) (FAHI+KS) questionnaire measures over time, accounting for clustering of responses within participants. There are three supplemental statements regarding participant perception of KS-specific symptoms: pain, swelling, and physical appearance. Agreement with each of these statements is graded using a Likert scale from 0 to 4. Responses to these statements may be dichotomized to reflect positive or negative impact of these symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Reid, MD, Principal Investigator — AIDS Malignancy Consortium
Locations (10):
- United States (10):
  - UC San Diego, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Street Clinic, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington